CLINICAL TRIAL: NCT03714542
Title: Prospective Evaluation of the Role of MRI in the Perioperative Management of Pancreas Adenocarcinomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, Professor, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-00108
Record Dates: First submitted 2016-08-05; First posted 2018-10-22 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pancreas Adenocarcinomas
MeSH Terms: interventions — Lead

ARMS (1):
- Pre- and postoperative MRI (Other): All patients will undergo a preoperative MRI and will have a postoperative follow-up with CT and MRI.
  Interventions: Other: Pre- and postoperative MRI

INTERVENTIONS:
Other: Pre- and postoperative MRI

SUMMARY:
The precision of MRI has improved over the past few years, in particular for the hepatobiliary and pancreatic pathologies. The role of MRI in the management of operated pancreas tumors remains nevertheless unclear and few studies have compared MRI to the actual gold standard (CT). Compared to CT, MRI is not only a morphologic imaging technique but also a functional imaging technique. MRI could therefore evaluate in a non-ionizing and dynamic way several important pre- and postoperative aspects after pancreaticoduodenectomy (PD). This study on the perioperative role of MRI includes 3 parts:

First, CT is known to minimize the real size of the pancreatic tumors and to underestimate the vascular invasion correlated to resectability. The preoperative determination of the resection surgical margins could be improved thanks to the high-contrast resolution of MRI.

Moreover, PD is a complex surgery encompassing a fragile anastomosis between the pancreatic parenchyma and the digestive tract. The permeability of the pancreatic anastomosis after PD remains presently unknown and has not been correlated to the clinical state of the patient. MRI associated with secretin injection allows evaluating this permeability, which cannot be done by CT due to the absence of functional evaluation.

Finally, present radiological follow-up after PD for tumors of the pancreatic head is performed with CT. The MRI performance has not been demonstrated yet in the context of follow-up. This imaging modality nevertheless offers unique specificities that are very interesting and that could be helpful for the diagnosis of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* indication for a PD for a resectable adenocarcinoma of the pancreatic head.

Exclusion Criteria:

* chronic pancreatitis
* absence of discernment
* patients not speaking French
* preoperative radio/chemotherapy
* patients with claustrophobia
* patients with metallic implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the MRI precision in the delimitation of circumferential resection margins | Preoperative MRI performed up to one month before the operation date.
  The preoperative MRI results will be compared to the anatomopathological results.

SECONDARY OUTCOMES:
Evaluation of the potential correlation between the tumor size and the resection margins. | Preoperative MRI performed up to one month before the operation date.
  The preoperative MRI results will be compared to the anatomopathological results. Tumor size and resection margins will be measured in cm.
Determination of the pancreatic anastomosis permeability | One year after the operation
  MRI with secretin injection
Determination of the rate of exocrine insufficiency | One year after the operation
  Elastase test in the stool
Correlation between anastomosis non-permeability and exocrine insufficiency. | One year after the operation
  Anastomosis non-permeability will be assessed with MRI with secretin one year after the operation. A score of permeability (number) will be appointed to determine permeability or not. Exocrine insufficiency will be defined by stool elastase measure <200 ug/g one year after the operation.
Evaluation of a questionnaire for pancreas exocrine insufficiency | One year after the operation
Evaluation of the MRI value to determine a recurrence in the follow-up of patients after PD | One year after the operation
  Comparison to the CT-scan

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospital, Lausanne, Canton of Vaud, Switzerland